CLINICAL TRIAL: NCT01556308
Title: Study of Inflammatory Mechanisms in Epidermolysis Bullosa Simplex- Dowling Meara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-AOI-02
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2012-03

CONDITIONS: Epidermolysis Bullosa Simplex Dowling Meara
Keywords: Dowling Meara; Epidermolysis bullosa; inflammation
MeSH Terms: conditions — Epidermolysis Bullosa; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DM-EBS (Experimental)
  Interventions: Procedure: Taking of liquid and top of blisters

INTERVENTIONS:
Procedure: Taking of liquid and top of blisters — the liquid and the top of blisters will be took.

SUMMARY:
Introduction: Epidermolysis Bullosa Simplex-Dowling-Meara (DM-EBS) is a rare genodermatosis characterized by spontaneous or post traumatic large cutaneous blisters. No curative treatment is actually available. Some data suggest a role of inflammation in the occurrence of blisters. The aim of this study is to study the epidermis inflammatory mechanisms in DM-EBS.

Material and methods: A first retrospective immunohistochemical study will be led on remainder skin biopsies of DM-EBS patients took for the diagnosis. A second clinical multicentric prospective study will be led on 8 patients older than 1 year with severe DM-EBS. After informed written consent, they will answer to a standardized questionnaire. In case of flare of the disease, the liquid and the top of the blisters will be took. Samples will be analyzed in the Pr Nicolas 851 INSERM unit. After centrifugation of the liquid blisters, the repartition of inflammatory cells will be evaluated by Fluorescence Activated Cell Sorting on the pellet. Markers of inflammation will be evaluated on the surnageant with Luminex® technical with a multiplex targeting cytokines and chemokines. An immuno-histochemic analysis in association with a quantitative PCR will be made on the top of the blisters. If unknown, genotypic study will be made.

Perspectives: A better comprehension of physiopathological mechanisms in DM-EBS could offer new therapeutic ways.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* older than 1 year-old
* severe Dowling Meara epidermolysis bullosa (more than 2 blisters per day)
* systematic written informed consent
* child consent
* affiliated to french social security

Exclusion Criteria:

* younger than one year-old
* no consent
* non affiliated to french social security
* participation to another clinical trial within 3 months ago
* intercurrent disease justifying the withdrawal of the study
* own patient decision to stop the study, withdrawal of informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Markers of inflammation in epidermis in patients with severe DM-BS | Baseline

SECONDARY OUTCOMES:
clinical characterization of DM-EBS Genotype-phenoty | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Archet 2, Nice, France